CLINICAL TRIAL: NCT00509210
Title: Study of Telaprevir in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VX06-950-012
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Hepatic Insufficiency
Keywords: Liver Disease
MeSH Terms: conditions — Hepatic Insufficiency; Liver Diseases | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: telaprevir (VX-950)

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of Telaprevir following administration of multiple oral doses to subjects with moderate and severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Child Pugh score of 7-9 or greater than 10
* Women of non-childbearing age

Exclusion Criteria:

* Tested positive for HIV, Hepatitis C, Hepatitis B

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Kwo, MD, Principal Investigator — Indiana University, Department of Medicine, Division of Gastroenterology/Hepatology
Locations (1):
- Indiana University, Department of Medicine,Division of Gastroenterology / Hepatology, Indianapolis, Indiana, United States